CLINICAL TRIAL: NCT04906681
Title: Implementation of a Rehabilitation Technology in Orthopedic and Neurological Rehabilitation to Increase Therapy Dosage: an Exploratory Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PXL University College (Other)
Collaborators: St-Trudo hospital, St-Truiden, Belgium (Unknown)
Responsible Party: Principal Investigator, Els Knippenberg, Principal investigator, PXL University College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exploration in St-Trudo
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Arthroplasty; Neurologic Disorder
Keywords: rehabilitation; technology
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arthroplasty, hip or knee (Experimental): Minimum 5x/week (of which minimal 3x/week with therapists and 2x/week during weekend), 30-60 minutes training, for 4 weeks, with i-ACT system. i-ACT provides individualised exercises based on patients own goalsetting.
  Interventions: Device: i-ACT
- Neurology: stroke or Parkinson disease (Experimental): Minimum 5x/week (of which minimal 3x/week with therapists and 2x/week during weekend), 30-60 minutes training, for 4 weeks, with i-ACT system. i-ACT provides individualised exercises based on patients own goalsetting.
  Interventions: Device: i-ACT

INTERVENTIONS:
Device: i-ACT — i-ACT is a Microsoft Kinect-based system that provides individualised exercises based on patients own goalsetting.

SUMMARY:
Rehabilitation technology is more and more implemented in conventional therapy to increase the dosage of therapy and/or increase patient's motivation towards therapy. In orthopedic as well as neurological rehabilitation it is important to exercise with enough intensity and repetitions to improve functional performance in activities of daily life, and consequently quality of life. At the moment, not all (rehabilitation) technologies are adapted towards the wishes and needs of both patients and therapists for everyday use in the clinical setting. Also, not all technologies are fit for independent use by the patients. Researcher of PXL have developed a Kinect-based system (i.e. i-ACT) for rehabilitation and performed supervised research with i-ACT in neurological and musculoskeletal rehabilitation, and older adults. Within this research, patients will exercise with i-ACT under supervision of their therapist during weekdays, but in the weekends they will be motivated by the medical staff to perform their exercises with i-ACT. The medical staff will be present for safety reasons, but the patient is asked to use and exercise with i-ACT as independent as possible. The aim of this research is to explore to which extend i-ACT is suitable for semi-independent use by patients in orthopedic or neurological rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* post-operation of arthroplasty (hip or knee), or official medical diagnosis of stroke or Parkinson's disease
* understand Dutch instructions
* patient at St-Trudo ziekenhuis
* experiencing problems in functional performance

Exclusion Criteria:

* neglect
* spasticity (Brunström Fugl-Meyer < 50)
* cognitive disfunction (Mini Mental State Examination < 24)
* visual impairment (blind, cataract, etc.)
* persons who are not able to exit electric wheelchair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline
  The Canadian Occupational Performance Measure (COPM) is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time. Scores range from 0 to 10 (best score) in each defined goal.
Canadian Occupational Performance Measure | 4 weeks
  The Canadian Occupational Performance Measure (COPM) is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time. Scores range from 0 to 10 (best score) in each defined goal.

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory | 1 week
  The Intrinsic Motivation Inventory (IMI) is a multidimensional measurement questionnaire intended to assess participants' subjective experience with, in this, i-ACT. The IMI consists of 6 subscales in which a person scores on a scale from 1 (totally not true) to 7 (totally true). Some scores need to be reversed by subtracting the response score from 8. A total IMI-score is not recommended, therefore subscale scores are used in the analyses. A higher score means a higher level of the aspect of the subscale.
Intrinsic Motivation Inventory | 4 weeks
  The Intrinsic Motivation Inventory (IMI) is a multidimensional measurement questionnaire intended to assess participants' subjective experience with, in this, i-ACT. The IMI consists of 6 subscales in which a person scores on a scale from 1 (totally not true) to 7 (totally true). Some scores need to be reversed by subtracting the response score from 8. A total IMI-score is not recommended, therefore subscale scores are used in the analyses. A higher score means a higher level of the aspect of the subscale.
System Usability Scale | 1 week
  Usability of a system, in this i-ACT. Range of scores from 0 (negative) to 100 (positive).
System Usability Scale | 4 weeks
  Usability of a system, in this i-ACT. Range of scores from 0 (negative) to 100 (positive).
Timed Up and Go test | Baseline
  The time between a person standing up from a chair, walking 3 meters before turning around and walking back to sit back in the chair.
Timed Up and Go test | 4 weeks
  The time between a person standing up from a chair, walking 3 meters before turning around and walking back to sit back in the chair.
2 Minute Walking Test | Baseline
  This is a measure of the distance a person can walk in 2 minutes.
2 Minute Walking Test | 4 weeks
  This is a measure of the distance a person can walk in 2 minutes.
Wolf Motor Function Test | Baseline
  Arm-hand functioning. The test contains 17 items and are scored from 0 (not able to perform tesk) to 5 (normal performance).
Wolf Motor Function Test | 4 weeks
  Arm-hand functioning. The test contains 17 items and are scored from 0 (not able to perform tesk) to 5 (normal performance).
Barthel Index | Baseline
  The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL. Scores range from 0 to 100.
Barthel Index | 4 weeks
  The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL. Scores range from 0 to 100.

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a possible publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 3 months after publication.